CLINICAL TRIAL: NCT07066137
Title: Motor Planning, Execution, and Modulation in Healthy Individuals and Patients With Movement Disorders or Neuromuscular Diseases Using Traditional Physical Activity or Advanced Devices to Enhance Motor Learning and Sensorimotor Processing
Brief Title: Motor Learning in Health and Movement Disorders: Role of Physical Activity and Advanced Devices
Acronym: Allena-mente
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Centro Neurolesi Bonino Pulejo (Other)
Responsible Party: Principal Investigator, Rocco Salvatore Calabrò, MED, PhD, IRCCS Centro Neurolesi Bonino Pulejo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Allena-mente
Record Dates: First submitted 2024-10-09; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Healthy Individuals (Controls); Parkinson Disease; Multiple Sclerosis; Alzheimer Disease; Dementia; Stroke
Keywords: Virtual Reality; motor rehabilitation; cognitive rehabilitation; Functional Recovery
MeSH Terms: conditions — Parkinson Disease; Multiple Sclerosis; Alzheimer Disease; Dementia; Stroke | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Type of Study: Interventional Objective: To evaluate the effects of advanced physiotherapy techniques and neuromodulation on motor and cognitive functions in both healthy individuals and patients with neurological conditions.
  Interventions: Physiotherapy, Cryotherapy, ultrasound therapy, laser therapy, music therapy, Neuromodulation: TMS, tDCS, Virtual Reality (CAREN) Proprioceptive stimulation and motor rehab, Intensive aerobic and anaerobic training.
  Groups:
  1. Healthy Participants
  2. Patients
  Phases:
  Recruitment: Initial evaluations and baseline data collection. Intervention: Application of treatments and regular assessments. Follow-up: Post-intervention evaluations and data analysis. Duration: Approximately 5 years. Outcome Measures: Improvements in motor performance, cognitive functions, and quality of life.
Who Masked: Investigator, Outcomes Assessor
Masking Description: In this study:
  Investigator: Not masked; investigators will be aware of the intervention each participant receives to monitor and administer the assigned treatments.
  Outcomes Assessor: Masked to the intervention each participant receives to ensure an unbiased evaluation of outcomes.
  Participants: Not masked; participants are aware of the intervention they are receiving as it involves different types of therapies and exercises.
  Data Analysts: Masked to participant group assignments during initial data analysis to prevent bias in interpreting results.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Healthy Subjects (Active Comparator): The subjects will undergo baseline examinations including MRI, spirometry, surface electromyography, 3D gait analysis, postural assessment and stabilometric analysis, O2 consumption measurement, neuropsychological assessment, ECG, and EEG.
  Subsequently, the healthy subjects (approximately 50) will undergo intensive aerobic and anaerobic training (including sensory-motor-cognitive training) and exercises on the CAREN platform. For the other 25 participants, transcranial magnetic stimulation (TMS)/transcranial direct current stimulation (tDCS) and music therapy will be added.
  Interventions: Other: Control group
- Experimental group (Experimental): As for the neurological patients (50), they will undergo posture and gait rehabilitation using the CAREN platform, while the other 25 will receive additional enhancement through non-invasive neuromodulation. This constitutes the other arm of the study.
  Interventions: Device: CAREN

INTERVENTIONS:
Device: CAREN — The interventions include proprioceptive stimuli combined with specific rehabilitation protocols, such as Tabata training, plyometric training, and visual-cognitive-motor enhancement with the S.V.T.A. method.
  Healthy subjects and athletes (about 50) will participate in intensive aerobic and anaerobic training, including sensory-motor-cognitive training and exercises on the CAREN platform. Another 25 participants will have TMS/tDCS and music therapy added to their regimen.
  Regarding neurological patients, 50 participants will undergo posture and gait rehabilitation using the CAREN platform, while 25 will receive non-invasive neuromodulation to enhance their rehabilitation outcomes. This arm of the study focuses on the recovery of motor and cognitive functions.
  This study uses the CAREN system as a tool for physical rehabilitation in neurological and healthy participants. The device is not being investigated for new indications and the study is conducted entirely in Italy.
  Arms: Experimental group
Other: Control group — the control group is typically the group that does not receive the experimental treatment or intervention, serving as a baseline to compare the effects of the intervention. However, in the context you're describing with healthy subjects and athletes, here's how it's structured:
  Healthy subjects and athletes (around 50 participants) will undergo:
  Intensive aerobic and anaerobic training Sensory-motor-cognitive training
  Additionally, 25 of these participants will receive:
  Transcranial Magnetic Stimulation (TMS) Transcranial Direct Current Stimulation (tDCS) Music therapy This approach allows for a comparison between the effects of the physical and cognitive training alone versus the enhanced effects when combined with neuromodulation (TMS, tDCS) and music therapy. This design will help in assessing the added value of these interventions on performance
  Arms: Healthy Subjects

SUMMARY:
The goal of this clinical trial is to investigate motor responses in healthy subjects and patients with movement disorders, brain and spinal cord injury, neuromuscular diseases, or cardiovascular diseases.

This study aims to evaluate the effectiveness of traditional physical activities combined with innovative interventions such as cryotherapy, ultrasound therapy, laser therapy, transcranial magnetic stimulation (TMS), and transcranial direct current stimulation (tDCS). It will also assess the impact of proprioceptive stimuli provided by either the immersive virtual reality (CAREN), or visuo-cognitive-motor enhancement (S.V.T.A.), and music therapy.

The main questions it aims to answer are:

How do these interventions affect motor activities and their functional recovery? What are the temporal and spatial changes in activation sequences related to motor learning and maintenance? When there is a comparison group: Researchers will compare outcomes between different intervention arms (e.g., physical activity with advanced devices vs. traditional methods) to find out if the advanced interventions result in better motor control and functional recovery.

Participants will:

* Undergo various rehabilitation protocols including physical activity and advanced interventions.
* Be assessed using different tool, such as fMRI, dtMRI, and NIRS to study in vivo neuroimaging and assess changes in brain function and connectivity.

DETAILED DESCRIPTION:
Objectives

Primary Objectives Investigating Motor Gesture Control: Study the sensory-motor structures and their connectivity in healthy participants and patients with neurological, cardiovascular, or neuromuscular conditions. This includes analyzing responses to advanced interventions such as transcranial magnetic stimulation (TMS), transcranial direct current stimulation (tDCS), and the CAREN (Computer Assisted Rehabilitation Environment) system.

Understanding Central Control Mechanisms: Assess spatial and temporal changes in brain activity during motor training and recovery processes, leveraging advanced neuroimaging techniques (e.g., fMRI, dtMRI, NIRS).

Secondary Objectives Postural Disorder Prevention: Develop strategies to enhance postural stability and prevent related disorders, improving sports performance and the quality of life in patients with neurodegenerative conditions.

Integration of Imaging and Psychometric Data: Employ multimodal data to uncover brain function patterns and inform rehabilitation strategies, contributing to personalized recovery protocols and optimized training methods.

Methodology Study Design

This is an interventional study aimed at evaluating the metabolic, functional, and neurophysiological aspects of motor responses in participants subjected to intensive physical and cognitive training. By combining traditional therapies with innovative technologies (e.g., CAREN, tDCS, TMS), the study will explore:

Central nervous system activation and connectivity. Temporal and spatial dynamics of motor learning and maintenance. The role of proprioceptive, visual, and auditory inputs in motor coordination.

Phases of Study Phase 1: Recruitment and Baseline Assessments Participants will be recruited through direct communication and provided with detailed study information.

Baseline evaluations will include:

Clinical and medical-sports assessment. Neuropsychological evaluation (e.g., MoCA, TMT, Stroop Test). Postural and gait analysis. Baseline imaging (MRI, EEG). Phase 2: Intervention and Data Collection

Participants will undergo structured interventions:

Physiotherapy sessions combined with neuromodulation techniques. Training on the CAREN system to assess and improve motor and postural functions.

Use of advanced devices for electromyographic data collection, oxygen consumption measurements, and 3D gait analysis.

Imaging and functional assessments will be repeated post-intervention.

Phase 3: Data Analysis and Dissemination Collected data will be anonymized, processed using advanced imaging and statistical algorithms, and analyzed for correlations between training responses and functional recovery.

Results will be published in high-impact international journals. Technologies and Assessments

Neuroimaging Techniques:

Functional and structural MRI (including T1-weighted, T2-weighted, and DTI sequences).

Analysis of mean diffusivity and fractional anisotropy to evaluate white matter integrity.

NIRS to assess cortical hemodynamics during tasks.

Neurophysiological Tools:

EEG and ECG to monitor the electrical activity of the brain and heart. Surface electromyography (EMG) to evaluate muscle activation patterns.

Advanced Rehabilitation Devices:

CAREN system: A virtual environment platform for motor and postural rehabilitation.

Alter-G/Gait Trainer 3 for assisted gait training. FLIR system for thermal imaging of muscular activity.

Neuropsychological Assessments:

Comprehensive cognitive evaluation, including MoCA, TMT, Stroop, and PASAT. Auditory anamnesis and visuomotor training (e.g., S.V.T.A.).

Population The study aims to recruit 150 participants, including healthy individuals and patients aged 18-60 years with neurological conditions (stroke, dementia, Parkinson's Disease, Multiple Sclerosis, Spinal Cord Injury). Detailed inclusion and exclusion criteria ensure the selection of suitable candidates.

Ethical and Administrative Aspects All participants will provide informed consent per ethical guidelines (Declaration of Helsinki and GDPR compliance).

The relevant Ethics Committee approves the study, with no additional costs or compensations.

Results will be transparently reported, adhering to international research standards.

ELIGIBILITY:
Inclusion Criteria:

* Montreal Cognitive Assessment (MoCA) score (adjusted for age and education) equal to or greater than 20.

Exclusion Criteria:

* Severe medical and psychiatric disorders potentially affecting the training

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2024-05-05 (Actual); Primary Completion 2026-05-05 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Amplitude of Motor-Related Event-Related Potentials (ERPs) During Gesture Execution Assessed by EEG. | Baseline (T0), post-intervention (T1, 12 weeks after baseline), and follow-up (T2, 3 months post-intervention).
  Motor-related EEG activity will be recorded during the execution of standardized gestures. The primary outcome is the mean amplitude (in µV) of specific ERP components (e.g., N200, P300) over motor cortex electrodes. Data will be averaged across trials for each participant and reported as group means ± standard deviation. Differences between healthy participants and clinical groups will be assessed using appropriate statistical tests.

SECONDARY OUTCOMES:
Respiratory Exchange Ratio (RER) During Submaximal Exercis | Baseline (T0), post-intervention (T1, 12 weeks after baseline), and follow-up (T2, 3 months post-intervention).
  Metabolic efficiency will be assessed through the respiratory exchange ratio (RER = VCO₂/VO₂) during submaximal steady-state exercise. RER will be measured at standardized workload levels and summarized as mean ± SD. Comparisons between groups or timepoints will assess changes in substrate utilization patterns.
Change in Global Cognitive Function as Measured by MoCA Total Score | Baseline (T0), post-intervention (T1, 12 weeks after baseline), and follow-up (T2, 3 months post-intervention).
  Cognitive function will be assessed using the Montreal Cognitive Assessment (MoCA). The primary outcome is the change in total score (range: 0-30) from baseline to post-intervention. Data will be summarized as mean ± SD and analyzed using paired or independent statistical tests, depending on the study design.

CONTACTS AND LOCATIONS:
Overall Officials: Rocco Salvatore Calabrò, PhD, Study Director — IRCCS Centro Neurolesi Bonino Pulejo
Locations (1):
- IRCCS Centro Neurolesi Bonino Pulejo, Messina, Italy/Me, Italy

IPD SHARING:
Plan to Share IPD: Yes
we plan to share individual participant data (IPD) with other researchers. The data will be made available through a secure platform, ensuring participant confidentiality and compliance with ethical guidelines. Access will be granted under a data use agreement that requires anonymization and outlines permitted uses. We encourage collaborative research and publication of findings derived from the shared data for a period of five years following the study's completion.
Supporting Information: SAP, CSR
Time Frame: Individual participant data (IPD) and supporting information will be available starting at the commencement of the study and will remain accessible for five years.
Access Criteria: Access to individual participant data (IPD) and supporting information will be granted to qualified researchers, including academic institutions, healthcare organizations, and other entities involved in neurorehabilitation research. Researchers will be able to access the anonymized IPD, study protocols, and relevant supporting information such as assessment measures and data collection methods. Access will be facilitated through a secure online data-sharing platform, where approved users can download the data after signing a data use agreement that outlines the terms of use and ensures compliance with ethical guidelines and participant confidentiality.
  This process aims to promote collaboration while safeguarding the integrity and privacy of the participants involved in the study.

REFERENCES:
- [Background] Bonanno M, De Pasquale P, De Marchis C, Lombardo Facciale A, Paladina G, Fonti B, Quartarone A, Calabro RS. Might patients with cerebellar ataxia benefit from the Computer Assisted Rehabilitation ENvironment (CAREN)? A pilot study focusing on gait and balance. Front Bioeng Biotechnol. 2024 Jun 24;12:1385280. doi: 10.3389/fbioe.2024.1385280. eCollection 2024. PMID 39011156